CLINICAL TRIAL: NCT07145554
Title: Comparative Effectiveness of Focal Extracorporeal Shock Wave Therapy and Steroid Injection in Piriformis Syndrome
Brief Title: f-ESWT vs Steroid Injection for Piriformis Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Hilal Busra Aycicek, MD, Specialist in Physical Medicine and Rehabilitation, Gulhane Training and Research Hospital
Other Study IDs: GulhaneTRH
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shock wave group
  Interventions: Other: Focal extracorporeal schock wave therapy
- Injection group
  Interventions: Procedure: Steroid Injection

INTERVENTIONS:
Other: Focal extracorporeal schock wave therapy — Participants in this group will receive a total of 5 sessions of focal extracorporeal shock wave therapy. Each session will deliver 1000 pulses per cm² to the affected piriformis muscle.
  Groups: Shock wave group
Procedure: Steroid Injection — Participants in this group will receive a single injection of corticosteroid into the piriformis muscle.
  Groups: Injection group

SUMMARY:
This study aims to compare two treatment methods for piriformis syndrome, a condition that can cause pain in the buttock and leg. Adult patients with piriformis syndrome will take part in the trial. Participants will be randomly assigned to one of two groups. One group will receive focal extracorporeal shock wave therapy (f-ESWT), a non-invasive treatment that uses sound waves. The other group will receive a steroid injection, which is a common treatment used to reduce pain and inflammation. The goal of this study is to find out which treatment is more effective in improving symptoms of piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with piriformis syndrome whose pain has persisted for three months or longer despite standard medical care and activity modifications.

Exclusion Criteria:

* Individuals with lumbar discopathy diagnosed by magnetic resonance imaging or electrodiagnostic study.
* Patients with coccyx pain.
* Individuals with mechanical or inflammatory disorders of the sacroiliac joint.
* Patients with pelvic region diseases.
* Pregnancy
* History of previous lumbar disc surgery.
* History of lumbar epidural block within the last 6 months.
* History of malignancy.
* Patients with signs of acute inflammation at the treatment site.
* Individuals with a cardiac pacemaker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with piriformis syndrome whose pain has persisted for three months or longer despite standard medical care. Participants include both men and women. Patients with lumbar discopathy, pelvic region diseases, sacroiliac joint disorders, pregnancy, previous lumbar disc surgery, recent lumbar epidural block, malignancy, acute inflammation at the treatment site, or cardiac pacemakers are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured by Numeric Rating Scale (NRS) | Baseline, 1 week, 4 weeks, and 12 weeks post-treatment
Quality of life measured by SF-36 questionnaire | Baseline and 4 weeks post-treatment